CLINICAL TRIAL: NCT03047915
Title: The Effects of a Music Intervention on Older Adults in the Emergency Department
Brief Title: Music in the Emergency Department (ED)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AAAQ3016
Record Dates: First submitted 2016-12-02; First posted 2017-02-09 (Estimated); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Anxiety
Keywords: Anxiety; Music intervention; Emergency department (ED)
MeSH Terms: conditions — Anxiety Disorders; Emergencies | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): All subjects enrolled will respond to questions assessing anxiety using the State Trait Anxiety Inventory (STAI), and pain using a 1-10 numerical score, and will have blood pressure and heart rate taken. Subjects randomized to the control group will continue the ED visit as usual.
- Music Group (Experimental): All subjects enrolled will respond to questions assessing anxiety using the State Trait Anxiety Inventory (STAI), and pain using a 1-10 numerical score, and will have blood pressure and heart rate taken. Subjects who are randomized to receive a music-listening intervention will listen to a choice of music for 30 to 60 minutes on a loaned iPad with disposable headphones. An hour after enrollment, participants will be asked the same questions assessing anxiety and pain, and will also have blood pressure and heart rate taken again.
  Interventions: Other: Music

INTERVENTIONS:
Other: Music — The intervention consists of listening to a choice of music for 30 to 60 minutes on a loaned iPad with disposable headphones.
  Arms: Music Group

SUMMARY:
This will be a randomized controlled study evaluating the effect of a music-listening intervention compared to standard care (control) during patient visit to the emergency department (ED). Randomization will be done with consecutive sealed envelopes.

Data collection will be prospective with administration of the State Trait Anxiety Inventory and collection of physiologic parameters (pain level, heart rate, blood pressure). Retrospective data will also be collected for covariate analysis (age, race/ethnicity, emergency severity index (ESI), pain medications administered during the ED visit, pain scores throughout ED visit, chief complaint, and ED discharge diagnosis).

DETAILED DESCRIPTION:
A visit to the emergency department (ED) is anxiety provoking for patients by nature. Contributing factors may include the sudden timing of the visit, a noisy environment, and waiting in anticipation of a serious diagnosis or bad news. Studies suggest that nearly 75% of adult ED patients may experience mild to severe anxiety in relation to the ED visit, but not directly related to their chief complaint. Anxiety can have deleterious effects on a patient in the clinical setting. Patients may report excessive pain complaints and manifest the typical signs and symptoms of anxiety (e.g. anorexia, dry mouth, nausea, chest pain), which can complicate diagnosis. Patient anxiety can also impose barriers to communication with ED staff, hindering successful delivery of important medical information. A visit to the ED may be particularly distressing for older adults (age 65+), for they are more likely than younger adults to have a greater ED length of stay before discharge home, receive more diagnostic tests and venipuncture for intravenous (IV) access, and have poorer pain care. Music listening as an anxiolytic has been shown to be effective across a variety of clinical settings, however there is a relative paucity of published data on the use of music listening for adult patients in the ED. No published studies, to the investigators' knowledge, have evaluated the effect of music listening on older adults in the ED.

ELIGIBILITY:
Inclusion Criteria:

* Present to the ED
* Aged 65 or over
* Speak English or Spanish

Exclusion Criteria:

* Individuals who are deaf
* Prisoners
* Individuals who cannot give informed consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 169 (Actual)
Dates: Start 2016-06; Primary Completion 2017-10 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Mean Change in STAI Score | Baseline and 1 hour post-intervention
  The STAI is scored from least/no anxiety (20 points) to severe anxiety (80 points). The mean change in STAI scores from before the intervention to after the intervention will be calculated by subtracting the first score from second score.

SECONDARY OUTCOMES:
Mean Change in Heart Rate (HR) | Baseline and 1 hour post-intervention
  The HR of patients will be recorded before and immediately after the intervention (for control subjects, 1 hour after enrollment). Difference in HR will be calculated by comparing pre to post and mean change calculated for each group.
Mean Change in Blood Pressure (BP) | Baseline and 1 hour post-intervention
  The BPs of subjects will be collected before and after the intervention (for control group, 1 hour after enrollment). Change in BP will be calculated per patient and the mean change calculated for each group.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen D. Sano, DO, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided